CLINICAL TRIAL: NCT01758848
Title: Physical Therapy for Overactive Bladder
Status: Terminated | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812091R
Record Dates: First submitted 2010-11-22; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; pelvic floor muscles; deep abdominal muscles
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Overactive bladder is a syndrome of symptoms. The core symptom is urgency with/without urge incontinence, frequency, nocturia. The prevalence of overactive bladder increased with age. The elderly is increasing with time, so the people who suffering from overactive bladder is also increasing. Research related to overactive bladder in the field of physical therapy is remained needed. The purposes of this study are to investigate the application of physical therapy to women with overactive bladder, emphasizing on the effect of voluntary muscle contraction for urgency inhibition, including the urodynamic study and clinical study.

There are three stages in this study. In the first stage, we are going to develop a specific health-related quality of life questionnaire for urinary incontinence in Taiwan version. One hundred and fifty women with urinary incontinence and fifty healthy women without lower urinary tract symptom will be recruited in the first year to investigate the reliability and validity of the questionnaire. The Short-Form 36, Chinese version, will be used as gold standard for validity. Fifty women with urgency will be recruited in the second stage to test the effect of muscle active contraction strategies to inhibit detrusor pressure and urgency. The three muscle active contraction strategies include pelvic floor muscle strong contraction, pelvic floor muscle tonic contraction, and transversus abdominis tonic contraction. The outcome variables including detrusor pressure of the urodynamic parameter and self-reported urgency score. Simultaneous image record by abdominal ultrasound during the urodynamic examination will be used to ensure the accuracy of muscle action. The predictors of success of strategy from the result of the second year will be used to stratify the patients in the third stage. Eighty women with urgency will be recruited in the final stage to examine the clinical effect of strategy for urgency inhibition.

DETAILED DESCRIPTION:
Overactive bladder is a syndrome of symptoms. The core symptom is urgency with/without urge incontinence, frequency, nocturia. The prevalence of overactive bladder increased with age. The elderly is increasing with time, so the people who suffering from overactive bladder is also increasing. Research related to overactive bladder in the field of physical therapy is remained needed. The purposes of this study are to investigate the application of physical therapy to women with overactive bladder, emphasizing on the effect of voluntary muscle contraction for urgency inhibition, including the urodynamic study and clinical study.

There are three stages in this study. In the first stage, we are going to develop a specific health-related quality of life questionnaire for urinary incontinence in Taiwan version. One hundred and fifty women with urinary incontinence and fifty healthy women without lower urinary tract symptom will be recruited in the first year to investigate the reliability and validity of the questionnaire. The Short-Form 36, Chinese version, will be used as gold standard for validity. Fifty women with urgency will be recruited in the second stage to test the effect of muscle active contraction strategies to inhibit detrusor pressure and urgency. The three muscle active contraction strategies include pelvic floor muscle strong contraction, pelvic floor muscle tonic contraction, and transversus abdominis tonic contraction. The outcome variables including detrusor pressure of the urodynamic parameter and self-reported urgency score. Simultaneous image record by abdominal ultrasound during the urodynamic examination will be used to ensure the accuracy of muscle action. The predictors of success of strategy from the result of the second year will be used to stratify the patients in the third stage. Eighty women with urgency will be recruited in the final stage to examine the clinical effect of strategy for urgency inhibition.

ELIGIBILITY:
Inclusion Criteria:

* women with overactive bladder

Exclusion Criteria:

-

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with overactive bladder
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
urinary diary | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Yih Tsauo, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan